CLINICAL TRIAL: NCT02445053
Title: Observational Study of Outcomes in Cystic Fibrosis Patients With Selected Gating Mutations on a CFTR Allele (The VOCAL Study)
Acronym: VOCAL
Status: Completed | Type: Observational
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: VX14-770-116; 2014-002704-24 (EudraCT Number)
Record Dates: First submitted 2015-05-11; First posted 2015-05-15 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ivacaftor
  Other Names: Kalydeco, VX-770

SUMMARY:
To describe the effectiveness of Kalydeco® treatment in patients with cystic fibrosis (CF) who have 1 of 8 non G551D gating CFTR mutations (G178R, S549N, S549R, G551S, G1244E, S1251N, S1255P, or G1349D).

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed diagnosis of CF16
* At least 1 allele with 1 of the following CFTR mutations: G178R, S549N, S549R, G551S, G1244E, S1251N, S1255P, G1349D
* Six years of age or older on the date of signed (Informed Consent Form) ICF, and where appropriate, date of assent
* Signed ICFs and, where appropriate, signed Assent Form
* Able to understand the study requirements and comply with study data collection procedures

Exclusion Criteria:

* Previously exposed to Kalydeco, except currently treated patients who started Kalydeco treatment within 6 months of enrollment
* Currently enrolled in a Kalydeco interventional study or other interventional therapeutic clinical study directed at CFTR modulation
* History of organ transplantation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients with CF, age 6 years or older, who have 1 of the following CFTR mutations on at least 1 allele: G178R, S549N, S549R, G551S, G1244E, S1251N, S1255P, or G1349D
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Pulmonary exacerbations - Number of pulmonary exacerbations and duration of treatment for pulmonary exacerbations during Kalydeco treatment compared to the period before Kalydeco treatment | 48 Months
Respiratory Microbiology - Percentage of patients with cultures positive for Pseudomonas aeruginosa during Kalydeco treatment compared to the period before Kalydeco treatment | 48 Months
Respiratory Microbiology - Percentage of patients with cultures positive for bacteria other than Pseudomonas aeruginosa and for fungi during Kalydeco treatment compared to the period before Kalydeco treatment | 48 Months
FEV1: Absolute change in percent predicted FEV1 during Kalydeco treatment | 48 Months
Measures of nutritional status: Absolute change in weight, weight-for-age Z score, body mass index (BMI), and BMI-for-age Z-score during Kalydeco treatment | 48 Months
Comorbidities: Incidence and prevalence of comorbidities during Kalydeco treatment compared to the period before Kalydeco treatment | 48 Months
Mortality: Incidence and cause of deaths | 48 Months
Organ transplantation: Incidence and reason for organ transplantations | 48 Months

OTHER OUTCOMES:
To explore the effect of Kalydeco treatment on Health-Related Quality of Life (HRQoL) in patients with CF and in caregivers of pediatric patients enrolled in the study. | 48 Months

CONTACTS AND LOCATIONS:
Locations (14):
- Italy (6):
  - Bari
  - Messina
  - Milan
  - Naples
  - Potenza
  - Verona
- Netherlands (6):
  - The Hague, South Holland
  - Amsterdam
  - Gronningen
  - Heidelberglaan
  - Nijmegen
  - Rotterdam
- United Kingdom (2):
  - London, Greater London
  - Birmingham, West Midlands